CLINICAL TRIAL: NCT00870636
Title: Compassionate Use Pan-VEGF Blockade for the Treatment of ROP (Compassionate Use BLOCK-ROP) Trial
Brief Title: Use of Pan-vascular Endothelial Growth Factor Receptor (Pan-VEGF) Blockade for the Treatment of Retinopathy of Prematurity (ROP) (Compassionate Use BLOCK-ROP)
Status: No longer available | Type: Expanded Access
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Thomas Lee, Associate Professor of Ophthalmology Keck School of Medicine, Children's Hospital Los Angeles
Other Study IDs: CCI-09-00044
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Retinopathy of Prematurity
Keywords: Pan-Vascular Endothelial Growth Factor Blockade; Safety; ROP; Bevacizumab; Avastin
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Bevacizumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Bevacizumab (Avastin) — Dosage of 0.75mg/0.03ml intravitreal injectable, one time only.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to provide access to intravitreal injection of Avastin in high-risk infants who do not otherwise qualify for study NCT00702819, an investigational multi-site study examining Avastin use for retinopathy of prematurity.

DETAILED DESCRIPTION:
Retinopathy of Prematurity (ROP) is a leading cause of blindness in children in developed countries around the world, and an increasing cause of blindness in developing countries. The retina lines the inside of the eye. It functions as "film" within the camera which is the eye. When an infant is born prematurely, the vascular network necessary to nourish the retina has not fully developed. As a consequence, in some infants abnormal vessels proliferate instead of the normal ones - a condition known as ROP. The abnormal vessels carry scar tissue along with them, and may lead to retinal detachment and blindness if the eye is not treated. The Multicenter Trial of Cryotherapy for Retinopathy of Prematurity (CRYO-ROP) Study demonstrated that ablation of the peripheral avascular retina reduced the risk of poor structural and visual outcome due to retinal distortion or detachment in ROP (1980's). The ablated retina is not functional and is not amenable to regeneration. Peripheral retinal ablation is not universally effective in fostering regression of ROP. This is particularly true for an aggressive form of ROP (aggressive posterior ROP, or APROP) which typically afflicts profoundly premature and infirm neonates. In this subset of infants, progression of ROP to bilateral retinal detachment and blindness occurs despite timely and complete peripheral retinal laser ablation.

The development of ROP is largely dependent on vascular endothelial growth factor (VEGF). When an infant is born prematurely the relatively hyperoxic environment the baby is introduced to shuts down the production of VEGF. Retinal maturation is delayed. Subsequently, at a time when intraocular VEGF levels would normally be declining late in the third trimester of pregnancy, abnormally high levels of VEGF are seen due to large areas of avascular retina and associated tissue hypoxia. The availability of FDA-approved drugs for anti-VEGF treatment renders it possible to treat such eyes off-label. Available drugs include pegaptanib sodium (Macugen) for partial blockage of VEGF-A, or drugs such as ranibizumab (Lucentis) and bevacizumab (Avastin), which cause complete blockage of VEGF-A. As VEGF is required in the developing retina for normal angiogenesis, our goal is not to penetrate tissue, but to block the excessive levels of VEGF trapped within the overlying vitreous which is responsible for the abnormal vasculature in ROP.

For purposes of this study we have chosen bevacizumab (Avastin), which will: a) attain complete blockage (vs. Macugen) of intravitreal VEGF-A, and; b) which is limited in its ability to penetrate tissues because it is a full antibody (vs. Lucentis, an antibody fragment specifically designed for better tissue penetration), and is more likely to restore VEGF homeostasis within the developing retina.

There is a nearly identical multi-site trial (NCT00702819) currently recruiting, which Childrens Hospital Los Angeles is a part of. However, that study has limiting enrollment criteria; this compassionate-use study was created to provide access to bevacizumab (Avastin) for high-risk infants who do not qualify for study NCT00702819.

ELIGIBILITY:
Inclusion Criteria:

* Inborn babies at CHLA NICU
* Outborn babies transferred to CHLA NICU
* Zone 1 or 2 ROP
* Adequate/appropriate laser ablation
* Failed standard laser treatment (persistent Plus disease at a minimum of 1 week post-laser)
* Post-menstrual age greater than 30 weeks

Exclusion Criteria:

* Zone 3 ROP
* Inadequate initial laser treatment
* Most recent laser treatment less than 1 week
* Evidence of tractional retinal detachment (exudative retinal detachment may be included in study group)
* Post-menstrual age less than 30 weeks
* Health not allowing for full protocol participation (determined by neonatologist)

Min Age: 30 Weeks | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lee, M.D., Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States